CLINICAL TRIAL: NCT00813163
Title: A Phase II Study of PEP02 as a Second Line Therapy for Patients With Metastatic Pancreatic Cancer
Brief Title: Study of PEP02 as a Second Line Therapy for Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PharmaEngine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEP0208
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Pancreatic Neoplasms
Keywords: Phase II study; Second line; Pancreatic cancer; Metastatic
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PEP02 (Experimental): Liposome Irinotecan
  Interventions: Drug: PEP02

INTERVENTIONS:
Drug: PEP02 — 120 mg/m2, IV infusion for 90 minutes on day 1 of each 21 days as a treatment cycle.
  Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: Liposome irinotecan

SUMMARY:
The purpose of this study is to see the effect of PEP02 in the treatment of metastatic pancreatic cancer.

DETAILED DESCRIPTION:
Gemcitabine monotherapy or a gemcitabine-based combination regimen is the standard first line therapy for advanced pancreatic cancer. After disease progression, there is no standard treatment available. In animal studies and a previous phase I trial, PEP02 has shown anti-tumor activity and preliminary efficacy in pancreatic cancer. In addition, a phase II study of free-form irinotecan single agent has already shown encouraging activity as second-line treatment for patients with advanced pancreatic cancer refractory to gemcitabine. The liposome formulation of PEP02 theoretically has therapeutic advantages over free-form irinotecan, such as site-specific delivery and extended release of drug. Hence PEP02 may be able to provide better efficacy than free-form irinotecan.

The primary purpose of this phase II study is to evaluate the activity of PEP02 as a second-line therapy in patients with metastatic pancreatic cancer failed to gemcitabine treatment. The primary goal is to measure the 3-month survival rate. An optimal Simon's 2-stage design will be used for this exploratory phase II study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of exocrine pancreas
* Metastatic disease
* Documented disease progression after treatment with 1 line of prior gemcitabine-based regimen
* Karnofsky performance status equal or more than 70

Exclusion Criteria:

* With active CNS metastases
* With clinically significant gastrointestinal disorder (e.g., bleeding, inflammation, occlusion, or diarrhea > grade 1)
* Major surgery or radiotherapy within 4 weeks
* Prior participation in any investigational drug study within 4 weeks
* With prior irinotecan treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Survival Rate | 3-month
  Survival rate at 3 months

SECONDARY OUTCOMES:
other efficacy endpoints | 6-8 weeks
  objective tumor response, PFS, duration of response, overall survival, tumor marker response of CA19-9, clinical benefit response
toxicities | 36 months
  All adverse events
pharmacogenetics | 24 months
  UGT1A1 polymorphism

CONTACTS AND LOCATIONS:
Overall Officials: Li-Tzong Chen, M.D., Principal Investigator — National Health Research Institutes, Taiwan; Andrew H Ko, M.D., Principal Investigator — University of California, San Francisco; Yu-Lin Lin, M.D., Principal Investigator — National Taiwan University Hospital
Locations (3):
- Comprehensive Cancer Center, UCSF, San Francisco, California, United States
- Taiwan (2):
  - National Health Research Institutes/National Chen-Kung Uiversity Hospital, Tainan
  - National Taiwan University Hospital, Taipei

REFERENCES:
- [Derived] Ko AH, Tempero MA, Shan YS, Su WC, Lin YL, Dito E, Ong A, Wang YW, Yeh CG, Chen LT. A multinational phase 2 study of nanoliposomal irinotecan sucrosofate (PEP02, MM-398) for patients with gemcitabine-refractory metastatic pancreatic cancer. Br J Cancer. 2013 Aug 20;109(4):920-5. doi: 10.1038/bjc.2013.408. Epub 2013 Jul 23. PMID 23880820